CLINICAL TRIAL: NCT06960577
Title: A Phase IIIb, Open-label, Single-arm, Global Study of Perioperative Durvalumab With Neoadjuvant ddMVAC or Gem/Cis in Patients With Muscle-invasive Bladder Cancer (NIAGARA-2)
Brief Title: Perioperative Durvalumab With Neoadjuvant ddMVAC or Gemcitabine/Cisplatin in Patients With Muscle-invasive Bladder Cancer (NIAGARA-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D933RC00002
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms; Immune Checkpoint Inhibitors; Methotrexate; Vinblastine; Doxorubicin; Cisplatin; Gemcitabine
Keywords: Muscle-invasive Bladder Cancer; Bladder Cancer; Immunotherapy; Durvalumab; Perioperative Durvalumab; ddMVAC; Gemcitabine; Cisplatin
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; Methotrexate; Vinblastine; Doxorubicin; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ddMVAC cohort (Experimental): Durvalumab + chemotherapy
  Interventions: Drug: Durvalumab; Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin
- gem/cis cohort (Experimental): Durvalumab + chemotherapy
  Interventions: Drug: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Durvalumab — Anti- PD-L1 Antibody.
  Arms: ddMVAC cohort
Drug: Methotrexate — Chemotherapy agent.
  Arms: ddMVAC cohort
Drug: Vinblastine — Chemotherapy agent
  Arms: ddMVAC cohort
Drug: Doxorubicin — Chemotherapy agent
  Arms: ddMVAC cohort
Drug: Cisplatin — Chemotherapy agent
  Arms: ddMVAC cohort
Drug: Durvalumab — Anti- PD-L1 Antibody
  Arms: gem/cis cohort
Drug: Gemcitabine — Chemotherapy agent
  Arms: gem/cis cohort
Drug: Cisplatin — Chemotherapy agent
  Arms: gem/cis cohort

SUMMARY:
The Phase IIIb NIAGARA-2 study aims to expand on the data from the Phase III NIAGARA study by investigating perioperative durvalumab in combination with investigator-selected cisplatin-based neoadjuvant chemotherapy (either ddMVAC or gemcitabine/cisplatin) in a clinical practice setting.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Participants with clinical tumour stage T2-T4aN0/1M0 or T1N1M0 with transitional or mixed transitional cell histology
* Patients must be planning to undergo radical cystectomy
* Patients who have not received prior systemic chemotherapy or immunotherapy for treatment of muscle-invasive bladder cancer
* ECOG performance status of 0 or 1
* Minimum life expectancy of 12 weeks at first dose of study medication

Exclusion criteria:

* Evidence of lymph node (N2-N3) or metastatic (M1) disease
* Inoperable tumour(s) with fixation to the pelvic wall on clinical examination
* Prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD 1, anti-PD L1 and anti-PD-L2 antibodies, excluding Bacillus Calmette-Guérin
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab
* Any concomitant medication known to be contraindicated to the chemotherapy (ddMVAC or gem/cis).
* Uncontrolled intercurrent illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
The safety of neoadjuvant durvalumab combined with ddMVAC or gem/cis prior to radical cystectomy (RC). | Up to 6 months
  Incidence of Grade 3 or 4 [possibly treatment-related adverse events (PRAEs)] as observed prior to RC.

SECONDARY OUTCOMES:
The safety and tolerability of perioperative durvalumab combined with ddMVAC or gem/cis. | Up to 2 years
  Incidence, severity, nature, seriousness, intervention/treatment, outcome, and causality of treatment-emergent adverse events, including PRAEs, adverse events of special interest, immune-mediated adverse events, adverse events (AEs), and serious adverse events; AEs resulting in study treatment interruption and discontinuation; laboratory findings.
The efficacy of perioperative durvalumab combined with ddMVAC or gem/cis in terms of event-free survival (EFS). | Up to 3 years
  EFS is defined as the time from first neoadjuvant durvalumab + chemotherapy treatment until the earliest occurrence of any of the following events:
  * First recurrence of disease after RC
  * First documented progression in participants who were medically precluded from RC
  * Time of expected surgery in participants who refuse to undergo RC or failure to undergo RC in participants with residual disease
  * Death due to any cause.
The efficacy of perioperative durvalumab combined with ddMVAC or gem/cis in terms of disease-free survival (DFS). | Up to 3 years
  DFS is defined as the time from the date of RC to the earliest of the first recurrence of disease post RC or death due to any cause.
The efficacy of perioperative durvalumab combined with ddMVAC or gem/cis in terms of OS. | Up to 3 years
  OS is defined as the time from first neoadjuvant durvalumab + chemotherapy until death due to any cause.
The efficacy of neoadjuvant durvalumab combined with ddMVAC or gem/cis followed by RC in terms of pathologic complete response (pCR). | Up to 3 years
  pCR rate is defined as the proportion of participants whose pathologic staging is T0N0M0 as assessed per local pathology review using specimens obtained via RC.
The efficacy of neoadjuvant durvalumab combined with ddMVAC or gem/cis followed by RC in terms of pathologic downstaging (pDS). | Up to 3 years
  pDS rate is defined as the proportion of participants whose pathologic staging is <P2 per local pathology review using specimens obtained via RC.

CONTACTS AND LOCATIONS:
Locations (53):
- Australia (9):
  - Research Site, Chermside
  - Research Site, Elizabeth Vale
  - Research Site, Heidelberg
  - Research Site, Hong Kong
  - Research Site, Kogarah
  - Research Site, Macquarie University
  - Research Site, Murdoch
  - Research Site, Port Macquarie
  - Research Site, St Leonards
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Jaú
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- France (18):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Chambray-lès-Tours
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Quint-Fonsegrives
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Suresnes
- Italy (3):
  - Research Site, Florence
  - Research Site, Orbassano
  - Research Site, Roma
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/